CLINICAL TRIAL: NCT02334020
Title: Effectiveness of Mental Health First-Aid Training in Denmark. A Randomized Controlled Trial With a Six-Month Follow-Up Supplemented With a Qualitative Study
Brief Title: Investigating the Impact of the Mental Health First-Aid Training Course in Danish Employees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Collaborators: TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Merete Nordentoft, Professor, Dr. Med Sc., Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MHFA Evaluation
Record Dates: First submitted 2014-12-08; First posted 2015-01-08 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Mental Health Impairment
Keywords: Mental illness; training; support; Mental Health
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training course (Experimental): 12 hour training course in Mental Health First-aid
  Interventions: Other: Mental Health First-aid
- Waiting list (Other): Waiting list design, hence delayed offering of Mental Health First-aid
  Interventions: Other: Mental Health First-aid

INTERVENTIONS:
Other: Mental Health First-aid — 2 days training course providing information on severe mental illness, in order to make people able to support in situations of crisis

SUMMARY:
The purpose of the study is evaluate the effect of the Mental Health First-aid training course on a Danish population of employees.

DETAILED DESCRIPTION:
Background:

Studies show a high and growing prevalence of mental disorders in the population worldwide. 25 % of the general population in Europe will during their lifetime experience symptoms related to a mental disorder. The Mental Health First Aid concept (MHFA) was founded in 2000 in Australia by Kitchener and Jorm, in order to provide the population with mental health first aid skills.

Objective:

The aim of the concept is, through an educational intervention (course), to increase confidence in how to help people suffering from mental health problems. Further, secondary aims are to increase the mental health literacy of the public by increasing knowledge, reduce stigma and initiate more supportive actions leading towards professional help. An investigation of the effect of MHFA offered a Danish population is needed.

Design and Methods:

The design is a randomized controlled superiority trial, in which 500 participants will be allocated to either the intervention group or the control group. The control group will attend the course six months later, hence waiting list design. From fall 2013 to spring 2014 participants will be educated in Mental Health First-aid following a manualized, two days MHFA course. All the participants will answer a questionnaire at base-line and at 6 months follow-up. The questionnaire is a back-translation of the questionnaire used in Australian trials. The trial will be complemented by a qualitative study, in which focus groups will be carried out.

Outcome:

The primary outcome measure is increased confidence in help-giving behavior among the participants. Secondary outcome will be increased knowledge of and improved positive attitudes towards people suffering from a mental health problem.

ELIGIBILITY:
Inclusion Criteria:

people, who in their line of work are in contact with many different individuals

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 538 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Increased confidence in help-giving behaviour as measured by comparing the intervention group after having attended the training course with the control group. (questionnaire) | 6 months
  Continuous outcome measures will be analyzed using generalized linear models and dichotomous outcome measures will be analyzed using binary logistic regression. Data will be analysed using IBM SPSS version 22.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Nordentoft, Prof. Dr.med, Principal Investigator — Mental Health Centre, in the capital region of Denmark
Locations (1):
- Mental Health Center Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Richardson R, Dale HE, Robertson L, Meader N, Wellby G, McMillan D, Churchill R. Mental Health First Aid as a tool for improving mental health and well-being. Cochrane Database Syst Rev. 2023 Aug 22;8(8):CD013127. doi: 10.1002/14651858.CD013127.pub2. PMID 37606172
- [Derived] Jensen KB, Morthorst BR, Vendsborg PB, Hjorthoj C, Nordentoft M. Effectiveness of Mental Health First Aid training in Denmark: a randomized trial in waitlist design. Soc Psychiatry Psychiatr Epidemiol. 2016 Apr;51(4):597-606. doi: 10.1007/s00127-016-1176-9. Epub 2016 Feb 2. PMID 26837214
- [Derived] Jensen KB, Morthorst BR, Vendsborg PB, Hjorthoj CR, Nordentoft M. The effect of the mental health first-aid training course offered employees in Denmark: study protocol for a randomized waitlist-controlled superiority trial mixed with a qualitative study. BMC Psychiatry. 2015 Apr 14;15:80. doi: 10.1186/s12888-015-0466-1. PMID 25884517